CLINICAL TRIAL: NCT05928091
Title: Evaluation of the Impact of an Expert Opinion During the Management of Patients With Severe Bleeding on Oral Anticoagulants.
Acronym: BANET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC IR 2019 BANET; 2021-A01684-37 (Other: ANSM)
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Hemorrhage
Keywords: anticoagulants; hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Centers will be randomized in two arms :
  * control group : each center will manage hemorrhage of participation as they usually did
  * interventional group : management of hemorrhage will be guided by the expert team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Doctors will manage bleeding as usual.
- Experimental group (Experimental): Investigators will call a phone number, and an expert will guide them to manage the bleeding.
  Interventions: Other: Phone call to an expert team

INTERVENTIONS:
Other: Phone call to an expert team — Patients will be treated as the expert said when the investigator called him
  Arms: Experimental group

SUMMARY:
The goal of this randomized clinical trial is to evaluate the impact of an expert opinion during the management of patients with severe bleeding on oral anticoagulants. The main question it aims to answer is :

• Does an expert help of decision during the management of patients with severe bleeding is superior to classic management ? The centers will be randomized in one of the two groups : control group and interventional group.

Patients will be followed for 3 months. At their inclusion they will be managed in conformity of the randomisation of their center.

They will be followed at hour 0 + 6 , H0+24 and at the end of hospitalization. After 3 months, they will be called to assess the occurrence of thrombotic events ou hemorrhage complications.

Researchers will compare the classic management versus the management with an expert opinion to see if the expert opinion is superior to classic management.

ELIGIBILITY:
Inclusion Criteria:

* Major patient treated with oral anticoagulants, admitted in an emergency department
* For suspected major bleeding defined according to the criteria of the International Society of Thrombosis and Haemostasis
* Able to give informed consent to participate in research or, in the event of an emergency, to take charge of a reference person
* Affiliated to a Social Security scheme.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient under guardianship, curatorship or safeguard of justice
* Administration within the last 24 hours of parenteral anticoagulant.
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of bleeding management | Hour 24
  The effectiveness of the management of bleeding will be evaluated with a rate of compliance with the recommendations in the event of major bleeding under oral anticoagulants

SECONDARY OUTCOMES:
Mortality rate all causes | Inclusion + 3 months
  Mortality rate all causes after 3 months
Hemostatic efficacy rate | Hour 24
  Hemostatic efficacy rate at 24 hours evaluated by an independent blinded evaluation committee
Specific mortality rate related to haemorrhage | Inclusion + 3 months
  Specific mortality rate related to haemorrhage after 3 months
Rate of new bleeding | Inclusion + 3 months
  Rate of new bleeding after 3 months
Thromboembolic events | Inclusion + 3 months
  Major thrombosis including symptomatic proximal venous thrombosis, symptomatic or non-symptomatic pulmonary embolism, ischemic vascular accident, myocardial infarction, cerebral thrombophlebitis, mesenteric portal thrombosis at 3 months
Duration of hospital stay | Inclusion + 3 months
  Duration of hospital stay over the entire 3-month follow-up
Changes in haemostasis values | Hour 6
  Rate of correction of haemostasis disorders at 6 hours post-reversion defined by an INR of less than 1.5 for Vitamin K Antagnist and normalization of activated partial thromboplastin time, prothrombin time, anti-Xa activity according to local normal values.
Rate of avoided and avoidable reversions | Hour 24
  Rate of avoided and avoidable reversions
Deadlines for implementing a reversion | Hour 24
  * Comparison of the time between the arrival of the patient in the emergency room and the implementation of the reversal
  * Comparison of the time between the patient's arrival in the emergency room and the performance of diagnostic imaging, particularly cerebral
  * Comparison of the time between the patient's arrival in the emergency room and the performance of a haemostatic procedure (interventional radiology, surgery, fibroscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Fares MOUSTAFA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (15):
- France (15):
  - CH Aurillac, Aurillac
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CH Le Puy, Le Puy-en-Velay
  - Hospice civils de Lyon, Lyon
  - CH de Montbrison, Montbrison
  - CH Montluçon, Montluçon
  - CH de Moulins, Moulins
  - CHU de Nice, Nice
  - CHR Orléans, Orléans
  - La Pitié-Salpétrière, Paris
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse
  - CHU Tours, Tours
  - CH de Vichy, Vichy